CLINICAL TRIAL: NCT00938171
Title: A Comparison of Local Anesthesia and General Anesthesia for Breast Cancer Surgery, a Prospective Randomized Trial
Brief Title: Comparing Local Anesthesia With General Anesthesia for Breast Cancer Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Yuan-Ching Chang MD, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MMH-I-S538; 97WHK0900049
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: Cytokine; Anesthesia; Local anesthesia; surgery; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anesthesia, Local; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local anesthesia (Active Comparator): local anesthesia with propofol sedation Target-controlled infusion (TCI) system will be used to maintain proper sedation level)
  Interventions: Procedure: Local anesthesia
- General anesthesia (Active Comparator): Patients receiving general anesthesia
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Local anesthesia — All patients will be then given adequate sedation with propofol and local anesthetic given by dermal infiltration in incision site and regional breast and axillary areas. The local anesthetic of choice will be 2 % lidocaine (Xylocaine) and 0.5% Bupivacaine (Marcaine) mixed with 7 % sodium bicarbonate and epinephrine (Bosmine)
  Other Names: LA
  Arms: local anesthesia
Procedure: General anesthesia — The method of general anesthesia for the GA group will be induced with fentanyl (1-2 μg/kg) and propofol (2.5 mg/kg). After placement of a laryngeal mask or endotracheal tube airway, anesthesia will be maintained with sevoflurane (end-tidal concentrations 1%-3%) in a 50% oxygen/nitrous oxide mixture.
  Other Names: GA
  Arms: General anesthesia

SUMMARY:
The purpose of this study is to determine therapeutic benefits by local anesthetic technique for breast cancer.

DETAILED DESCRIPTION:
Experimental and clinical studies have shown that surgical trauma and stress affects the immune system including both the innate and adaptive immune responses.

The break of immune homeostasis might enhance tumor growth and spread. Minimal invasive surgical procedures have been shown to be beneficial to patients in terms of preserving better systemic immune function. Impaired cellular immunity after general anesthesia has significant undesirable effects on tumor surveillance after breast surgery. The local block technique might avoid the surgery inducing neuroendocrine, metabolic, and cytokine responses, which will offer some advantages from better preservation of early postoperative cellular immune function and attenuate disturbance in the inflammatory mediators. Our research will focus on the effects of local block anesthesia on mediators that may be important in inflammatory response, tumor cell dissemination, deposition, and propagation in the early postoperative period. As importantly, local block method is not only a safe procedure but also reduces the need for post operative opioids and prevents nausea following breast cancer which can result in markedly reduced hospital stay and health costs. It is plausible that inhibition of the surgical responses by local block anesthesia may attenuate perioperative tumor enhancing factors and/or potential beneficial actions of lidocaine infiltration combined with propofol sedation per se in anticancer effect to have better cancer control.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven breast cancer Scheduled for mastectomy and axillary node dissection in a single procedure.

Exclusion Criteria:

* previous surgery within the preceding 2 wk those other than ASA physical status I or II any contraindication to either local anesthesia or opioid analgesia

Ages: 21 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain scores | Until PACU discharge and for 24 hours

SECONDARY OUTCOMES:
disease free survival | 5 years
Episodes of nausea or vomiting | 24 hours
Overall patient satisfaction | After hospital discharge and six months later
The need for postoperative opioids | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: YuanChing Chang, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay memorial hospital, Taipei, Taiwan